CLINICAL TRIAL: NCT02139956
Title: Ultrasonic Assessment of the Urethra and the Vagina in Normal Continent Women and Women Suffering From Stress Urinary Incontinence
Brief Title: Assessment of the Internal Urethral Sphincter and the Vagina by Three Dimensional Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, dr mervat ekky, mekky, Ain Shams University
Other Study IDs: mekky
Record Dates: First submitted 2014-05-06; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Urinary Incontinence Due to Urethral Sphincter Incompetence
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days

GROUPS / COHORTS (2):
- stress urinary incontinence: group 1 women with stress urinary incontinence by ultrasonography
  Interventions: Device: ultrasonography
- continent group: group 2 women without stress urinary incontinence by ultrasonography
  Interventions: Device: ultrasonography

INTERVENTIONS:
Device: ultrasonography — open
  Other Names: vilson E6; transvaginal probe

SUMMARY:
Continent women have an intact internal urethral sphincter that extends from the bladder neck down to the perineal membrane. The internal urethral sphincter is a strong collagen muscle tissue cylinder lined by urothelium. On ultrasound scanning tissue echo will be detected torn internal urethral sphincter will not stand sudden rise of abdominal pressure. Three dimensional ultrasound assessment of the internal urethral sphincter is very sensitive and specific for the diagnosis of stress urinary incontinence.

DETAILED DESCRIPTION:
The internal urethral sphincter used to be said it's a muscular ring but the investigators will visualize by three dimensional ultrasound it's a cylinder in shape and it's the cause of stress urinary incontinence by being torn by stretching the vagina during normal delivery.

ELIGIBILITY:
Inclusion Criteria:

* signed an informed consent
* patient with stress urinary incontinence
* patient have done a vaginal delivery
* patient with genital prolapse

Exclusion Criteria:

* refusal to sign an informed consent
* patient have urinary tract infection
* patient with pregnancy
* patient have vaginal infection
* patient who has undiagnosed vaginal bleeding

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: out patient [clinics] and in patient
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
evaluation of the internal urethral sphincter and assesst the extend and degree of the torn internal urethral sphincter | 6 month
  we are going to do 3d ultrasound by transvaginal probe to see the internal urethral sphincter if torn or not and evaluate the morphology of the urethra and pelvic floor structure

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Result] Kruger JA, Dietz HP, Budgett SC, Dumoulin CL. Comparison between transperineal ultrasound and digital detection of levator ani trauma. Can we improve the odds? Neurourol Urodyn. 2014 Mar;33(3):307-11. doi: 10.1002/nau.22386. Epub 2013 Feb 22. PMID 23436235